CLINICAL TRIAL: NCT07189052
Title: Effects of a Virtual Reality-Based Rehabilitation Program on Pain and Function in Individuals With Chronic Neck Pain
Brief Title: Virtual Reality Program for Managing Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Hatice Çeitn, Asst.Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRTR34T
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neck Pain
Keywords: virtual reality; serious gaming; chronic; neck; pain; rehabilitation; conventional; technologic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: (1) virtual reality-based rehabilitation or (2) conventional therapy. Both groups will complete the same categories of therapeutic exercises (breathing, stretching, cervical range-of-motion, and posture-strengthening), but the VR group performs a gamified version in an immersive virtual environment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Treatment Group (Experimental): Participants in this group will receive a virtual reality-based rehabilitation program developed by the investigators for individuals with chronic neck pain. The program includes four structured components: (1) diaphragmatic breathing with guided head movements in a seaside setting; (2) stretching performed through avatar-controlled jet-ski tasks to collect targets; (3) cervical range-of-motion exercises covering flexion, extension, lateral flexion, and rotation; and (4) posture-strengthening tasks to promote scapular and postural control. All exercises correspond to conventional therapy content but are delivered as immersive, game-adapted tasks. The program will be delivered for 8 weeks, 2 sessions per week (16 sessions total), each lasting about 20 minutes.
  Interventions: Other: Virtual Reality Rehabilitation
- Conventional Therapy Group (Active Comparator): Participants in this group will receive a therapist-guided physiotherapy program for chronic neck pain. The program includes: (1) diaphragmatic breathing, 10 repetitions; (2) trapezius stretching (right and left), 10 repetitions of 15 seconds each; (3) cervical range-of-motion exercises (flexion, extension, lateral flexion, rotation), 10 repetitions of 5 seconds each; and (4) posture-strengthening with proprioceptive neuromuscular facilitation for scapular retraction, 3 sets of 10 repetitions. The program will be delivered for 8 weeks, 2 sessions per week (16 sessions total), each lasting about 20 minutes.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Virtual Reality Rehabilitation — A virtual reality-based rehabilitation program including breathing, stretching, cervical range-of-motion, and posture-strengthening tasks delivered in a gamified seaside environment using a head-mounted VR display. Sessions will last 20 minutes, performed twice per week for 8 weeks (16 sessions total) under supervision.
  Arms: Virtual Reality Treatment Group
Other: Conventional Rehabilitation — Standard physiotherapy including diaphragmatic breathing, trapezius stretching, cervical range-of-motion, and posture-strengthening with proprioceptive neuromuscular facilitation. Sessions will last 20 minutes, performed twice per week for 8 weeks (16 sessions total) under supervision.
  Arms: Conventional Therapy Group

SUMMARY:
The goal of this clinical trial is to find out if a virtual reality-based rehabilitation program developed by our team can help people with chronic neck pain.

The main questions it aims to answer are:

* Does the VR program reduce neck pain?
* Does it improve daily function and quality of life?

Participants will:

* Take part in a supervised virtual reality exercise program for 8 weeks, attending 3 sessions per week (24 sessions in total).
* Each session will last about 45 minutes.
* Complete tests and questionnaires about their pain, disability, and overall well-being before and after the program.

DETAILED DESCRIPTION:
This trial evaluates a virtual reality (VR)-based rehabilitation program developed by our team for people with chronic neck pain, compared against conventional therapy (CT) delivered as standard physiotherapy. Both programs share the same exercise components (breathing, stretching, range-of-motion, and posture-strengthening); the VR arm provides a game-adapted version in an immersive "beach and ocean" setting via a head-mounted display. Participants in both arms attend 20-minute sessions, twice per week over the intervention period. ￼ ￼

VR-Based Rehabilitation (Intervention)

The VR treatment module is structured into four components that run continuously within a beach-themed scenario:

* Breathing component: Before gameplay, participants are taught diaphragmatic breathing. In VR, the avatar starts on a deck chair by the sea; on-screen prompts guide the participant to inhale while lifting the head toward the sky and exhale while lowering toward the sand (approx. 5 minutes). ￼
* Stretching component: The avatar rides a jet-ski along the shoreline and the participant collects coins arranged bilaterally, promoting controlled neck movements within the stretching block. ￼
* Range-of-motion component: Therapeutic tasks cue cervical flexion, extension, lateral flexion (right/left), and rotation (right/left) as part of the game flow, mirroring the clinical ROM targets. ￼
* Posture-strengthening component: Gamified tasks reinforce postural and scapular control consistent with the conventional program's strengthening principles. ￼

Overall, the VR arm delivers the same exercise content as CT, but as a game-adapted version in an immersive beach setting via VR glasses. ￼

Conventional Therapy (Comparator)

The CT arm performs the same exercise categories as standard, therapist-guided physiotherapy with predefined sets/repetitions:

* Diaphragmatic breathing: 10 repetitions. ￼
* Stretching: Trapezius (right and left) - 10 repetitions × 15 seconds each side. ￼
* Neck ROM exercises: Flexion & extension; right/left lateral flexion; right/left rotation - 10 repetitions × 5 seconds per movement. ￼
* Posture-strengthening: Proprioceptive Neuromuscular Facilitation (PNF)-based scapular retraction - 3 sets × 10 repetitions (with facilitation at the start of each series). ￼

Dose & schedule: Both arms follow 20-minute sessions, twice weekly; outcomes (e.g., pain, disability, kinesiophobia, quality of life) are recorded pre-/post-intervention (detailed in the Outcomes section).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of chronic neck pain (≥ 6 months duration)
* Ability to participate in rehabilitation sessions
* Willingness to provide written informed consent

Exclusion Criteria:

* Previous adverse experience with virtual reality
* Photophobia (UPSIS-12 score > 12)
* Migraine (≥ 2 positive responses on ID-Migraine questionnaire)
* Presence of any neurological deficit
* History of spinal surgery
* Medical conditions interfering with participation, including orthopedic, inflammatory, cardiovascular, rheumatologic, or vestibular disorders
* Pregnancy
* Epilepsy or other neurological conditions causing photosensitivity
* Congenital spinal cord malformations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and at the end of the study.
  Pain severity will be measured using the Visual Analog Scale (VAS), a 10-cm line ranging from 0 (no pain) to 10 (worst imaginable pain), where participants indicate their average neck pain intensity over the past week. Higher scores represent greater pain (worse outcome).
Neck Disability | Baseline and at the end of the study.
  Functional disability will be evaluated using the Neck Disability Index (NDI), a 10-item self-report questionnaire assessing daily activities affected by neck pain. Each item is scored from 0 to 5, yielding a total score range of 0 (no disability) to 50 (maximum disability). Higher scores indicate greater disability (worse outcome).
Cervical Range of Motion | Baseline and at the end of the study.
  Cervical range of motion (flexion, extension, right/left lateral flexion, and right/left rotation) will be measured using the CROM device. Higher values indicate greater mobility.
Proprioception | Baseline and at the end of the study.
  Proprioceptive accuracy will be assessed by measuring joint position sense error in degrees using the CROM device. Higher error values indicate poorer position sense.

SECONDARY OUTCOMES:
Life Quality | Baseline and at the end of the study.
  Quality of life status will be measured using the Short Form-36 Health Survey (SF-36). Scores range from 0 (worst possible health status) to 100 (best possible health status). Higher scores indicate better health-related quality of life.
Kinesiophobia | Baseline and at the end of the study.
  Fear of movement will be assessed using the Tampa Scale of Kinesiophobia (TSK), a 17-item self-report questionnaire. Each item is scored from 1 to 4, yielding a total score range of 17 (no kinesiophobia) to 68 (maximum kinesiophobia). Higher scores indicate more severe kinesiophobia (worse outcome).
Treatment Adherence | At the end of the study.
  Attendance at scheduled sessions will be recorded to determine adherence to the VR or conventional therapy program. Higher percentages reflect better adherence.
Participant Satisfication | At the end of the study.
  Perceived overall change will be evaluated using the Global Perceived Effect (GPE) Scale, a 7-point Likert-type scale assessing the participant's impression of improvement following the treatment program. Scores range from 1 (much worse) to 7 (much better), with 4 indicating no change. Higher scores indicate greater perceived improvement (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Department of neurosurgery, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) because of privacy and confidentiality concerns.

REFERENCES:
- [Background] Ruf M, Welk T, Muller M, Merk HR, Harms J. Ventral cancellous bone augmentation of the dens and temporary instrumentation C1/C2 as a function-preserving option in the treatment of dens pseudarthrosis. J Spinal Disord Tech. 2010 Jun;23(4):285-92. doi: 10.1097/BSD.0b013e3181aac6ff. PMID 20110831